CLINICAL TRIAL: NCT07132411
Title: Talk With Me Baby: Leveraging Well-Child Care to Enhance the Early Home Language Environment
Acronym: TWMB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00151172; 5R01HD112446-02 (NIH)
Record Dates: First submitted 2025-07-02; First posted 2025-08-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Child Language; Language Delay; Developmental Milestones
Keywords: well-child care; primary care practices; home language environment; preventative intervention; language development; language promotion intervention
MeSH Terms: conditions — Language Development Disorders

STUDY DESIGN:
Intervention Model Description: A pragmatic type 1 hybrid effectiveness-implementation cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Talk With Me Baby Clinics (Experimental): In TWMB clinics, TWMB will be delivered within usual WCC workflows for anticipatory guidance during the clinical encounter. TWMB is delivered by the primary clinician (i.e., pediatrician/family medicine physician; physician assistant; nurse practitioner) and/or a clinician and care team. TWMB targets key evidence-based language promotion strategies that previous research has shown to improve child language outcomes. TWMB training involves didactic and practice-based instruction (CME/CNE) that includes: (a) a brief review of the science behind why language promotion matters; (b) focused instruction (with video examples and modeling) on how to deliver components of TWMB, including the TWMB Checklist and Language Nutrition Prescription; and (c) live practice and role play with the trainer on delivering TWMB across child ages and families.
  Interventions: Behavioral: Patients in Talk With Me Baby Clinics
- Care-As-Usual Clinics (Active Comparator): Providers/care teams will deliver care-as-usual WCC visits for all children. Parent-child participants in Control clinics will receive WCC anticipatory guidance care as usual. No treatment control is in line with the literature on randomized behavioral/educational interventions.
  Interventions: Behavioral: Patients in Care-As-Usual Clinics

INTERVENTIONS:
Behavioral: Patients in Talk With Me Baby Clinics — Parent-child participants in TWMB clinics will attend their regular WCC visits (scheduled per routine clinic processes) following the AAP Periodicity Schedule.
  Arms: Talk With Me Baby Clinics
Behavioral: Patients in Care-As-Usual Clinics — Parent-child participants in Care-As-Usual clinics will attend their regular WCC visits (scheduled per routine clinic processes) following the AAP Periodicity Schedule. Measures will be completed at five time points.
  Arms: Care-As-Usual Clinics

SUMMARY:
Language-rich interactions with a parent or caregiver can serve as a protective factor for young children, by supporting their language development and other positive long-term outcomes, but existing interventions have not had the necessary reach to families who need this information the most. This study utilizes the primary care setting as a low cost, scalable way to deliver language promotion intervention. Specifically, we will test the effectiveness and explore implementation of language promotion intervention (Talk With Me Baby) that embeds within anticipatory guidance during pediatric well-child care to boost early language development and optimize health, academic, and economic outcomes.

DETAILED DESCRIPTION:
The quality of early language interactions with parents and caregivers in early childhood has long-term implications for a child's social, economic, and physical heath. Differences in the home language environment (HLE) are well established and cross all sociodemographic characteristics. Although several decades of research have identified evidence-based strategies that enhance the HLE and improve child outcomes, they have failed to reduce population-level differences in child language development and long-term outcomes. The study utilizes Talk With Me Baby (TWMB) as a novel tool to increase language building interactions between parent/caregiver and child. Because TWMB is delivered in the primary care setting (which reaches up to 98% of families with infants and toddlers), it is scalable, low-cost, and universal. With TWMB, healthcare providers can embed evidence-based language promotion into their well-child care (WCC) anticipatory guidance for all children age 0-3 years. TWMB builds on decades of well-controlled language intervention efficacy trials and has been deployed clinically for 8+ years. This study is a type 1 hybrid effectiveness implementation trial to measure the impact of TWMB on gains in the HLE and subsequent child language outcomes. The trial is both randomized and controlled across 2 sites: a TWMB intervention group (8 clinics) and a care-as-usual control group (8 clinics). In TWMB clinics, providers and care teams will be trained to deliver TWMB during all 2-24 month WCC visits. Across TWMB and control clinics, we will enroll 25 parent-child dyads in each clinic (n=400 total) prior to their 2-month WCC visit and follow them through their 24-month WCC visit.

ELIGIBILITY:
Inclusion Criteria for Participants:

* Child must be enrolled prior to attending their 2-month WCC visit, age 1 month (+/- 30 days)
* Full term (>=37 weeks gestation)
* Singleton birth
* Home language of English and/or Spanish
* Child must receive WCC at a participating clinic

Exclusion Criteria for Participants:

* Child with a severe congenital disorder that would affect neurodevelopmental outcomes, or hearing impairment that could affect participation
* Parent does not live with or spend >=2 days/week with the child
* Family does not plan to continue services at the clinic

Inclusion Criteria for Clinics:

* A primary care practice (family medicine or pediatric model) that delivers WCC for children from 0-36 months old
* A minimum of 30% Medicaid/uninsured visits/year
* A minimum of 300 unique 0 to 36-month-old patients/year

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Change in parent language-promotion behavior | Child age 1, 6, 12, and 18 months old
  Change in parent language-promotion behavior (as measured by Language Environment Analysis [LENA] Conversational Turn Count) at each assessment time point (child age 1, 6, 12, and 18 months old) for parent-child dyads in TWMB clinics, compared to care-as-usual clinics.
Child total language | Child age 24 months old
  Child language (as measured by the Preschool Language Scale-5 [PLS-5/PLS-5 Spanish] for Total Language) at child age 24 months old for parent-child dyads in TWMB clinics, compared to care-as-usual clinics.
Child receptive language | Child age 24 months old
  Child receptive language (as measured by the Preschool Language Scale-5 [PLS-5/PLS-5 Spanish] for Receptive Language) at child age 24 months old for parent-child dyads in TWMB clinics, compared to care-as-usual clinics.
Child expressive language | Child age 24 months old
  Child expressive language (as measured by the Preschool Language Scale-5 [PLS-5/PLS-5 Spanish] for Expressive Language) at child age 24 months old for parent-child dyads in TWMB clinics, compared to care-as-usual clinics.

SECONDARY OUTCOMES:
Change in parent language promotion knowledge | Child age 1, 12, and 24 months old
  Parent language promotion knowledge (as measured using the Survey of Parent Expectations & Knowledge [SPEAK] total score) at each child age 1, 12, and 24 months old for parent-child dyads in TWMB clinics, compared to care-as-usual clinics.
Change in Child vocalizations and verbalizations | Child age 1, 6, 12, and 18 months old
  Change in child vocalizations and verbalizations (as measured by Language Environment Analysis [LENA] Child Vocalization Count percentile scores) at child age 1, 6, 12, and 18 months old for children in TWMB clinics, compared to care-as-usual clinics.
Change in child receptive vocabulary | Child age 12, 18, and 24 months old
  Change in child receptive vocabulary (as measured by MacArthur-Bates Communicative Development Inventories [MBCDI] Short Form and Spanish Inventario Short Form I/II) at child age 12, 18, and 24 months for children in TWMB clinics, compared to care-as-usual clinics.
Change in child expressive vocabulary | Child age 12, 18, and 24 months old
  Change in child expressive vocabulary (as measured by MacArthur-Bates Communicative Development Inventories [MBCDI] Short Form and Spanish Inventario Short Form I/II) at child age 12, 18, and 24 months for children in TWMB clinics, compared to care-as-usual clinics.
Parent contingent responding scores for a subset of the sample | Child age 18 months old
  Parent contingent responding scores (as measured by behavioral coding of home video recordings during daily routines) at child age 18 months for children in TWMB clinics, compared to care-as-usual clinics.
Parent contingent verbal scaffolding scores for a subset of the sample | Child age 18 months old
  Parent verbal scaffolding scores (as measured by behavioral coding of home video recordings during daily routines) at child age 18 months for children in TWMB clinics, compared to care-as-usual clinics.
Feasibility of intervention for treatment arm only | Upon study completion, approximately 2 years
  Feasibility of intervention (as assessed by the Feasibility of Intervention Measure [FIM]at post-intervention. The study team also plans to conduct interviews with the clinics with the highest and lowest FIM scores to identify facilitators and barriers to implementation.
Acceptability of intervention for treatment arm only | Upon study completion, approximately 2 years
  Acceptability of intervention (as assessed by the Acceptability of Intervention Measure [AIM]) at post-intervention. The study team also plans to conduct interviews with the clinics with the highest and lowest AIM scores to identify facilitators and barriers to implementation.
Appropriateness of intervention for treatment arm only | Upon study completion, approximately 2 years
  Appropriateness of intervention (as assessed by the Intervention Appropriateness Measure [IAM]) at post-intervention. The study team also plans to conduct interviews with the clinics with the highest and lowest IAM scores to identify facilitators and barriers to implementation.

OTHER OUTCOMES:
Moderator: Family strengths and parent resources | Child age 1 month old
  Family strengths and parent resources (as measured using the Healthy Families Parenting Inventory (HFPI) total score) at baseline.
Mediator: Parent language promotion knowledge | Child age 1 month old
  Parent language promotion knowledge (as measured using the Survey of Parent Expectations & Knowledge [SPEAK] total score) at baseline.
Mediator: Home language environment for child outcomes | Child age 1, 6, 12, and 18 months old
  Home language environment (HLE) as measured using Conversational Turns [CT percentile score] at each child age 1, 6, 12, and 18 months old.
Mediator: Dosage of parent input for child outcomes | Child age 1, 6, 12, and 18 months old
  Dosage of parent language input as measured using LENA Adult Word Count [AWC percentile score] at each child age 1, 6, 12, and 18 months old.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda J Salley, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol